CLINICAL TRIAL: NCT06731465
Title: Efficiency, Efficacy, Periodontal and Occlusal Outcomes for Clear Aligners Versus Pre-adjusted Orthodontic Appliances in Moderately Crowded Lower Incisor Treatment: a Randomized Clinical
Brief Title: Efficiency, Efficacy, Periodontal & Occlusal Outcomes for Aligners Versus Fixed Orthodontic Appliances in Crowded Incisor Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Mais Medhat Sadek AbdelAzim, Assistant Professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-23-05-13-01-PG
Record Dates: First submitted 2024-10-31; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Crowding of Anterior Mandibular Teeth
Keywords: Clinical trial; Clear Aligners; Fixed Pre-adjusted Edgewise Orthodontic Appliance; Orthodontic Treatment; Efficiency; Efficacy; Periodontal Outcomes; Randomized Clinical Trial; Orthodontic alignment time; Occlusal outcomes
MeSH Terms: interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: The interventional study model used in this study is a two-arm, parallel-group, randomized controlled trial (RCT) with a 1:1 allocation ratio between two treatment arms: clear aligners and fixed braces. The study is structured to evaluate the treatment efficiency, efficacy and periodontal as well as occlusal parameters in participants treated with fixed labial braces or clear aligners for alignment of moderately crowded lower incisors. Block randomization is used to ensure an equal number of participants in each group, reducing potential imbalances in group size and baseline characteristics. Both groups will have regular progress checks every 4-6weeks, with adjustments or new aligners provided based on treatment progression.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed labial braces group (Active Comparator): Participants in this group will be treated with pre-adjusted fixed orthodontic appliances.
  Interventions: Device: Fixed pre-adjusted edgewise orthodontic appliance
- Clear aligner group (Active Comparator): Participants in this group will receive clear aligners customized based on a digital model of each patient's dentition.
  Interventions: Device: Clear aligner therapy

INTERVENTIONS:
Device: Clear aligner therapy — Participants in this group will receive clear aligners (EON Aligner, Minneapolis), designed and customized based on a digital model of each patient's dental structure. Aligners will be worn for at least 22 hours daily, and patients will change to a new aligner depending on treatment progress.
  Other Names: Clear aligners; Clear aligner therapy (CAT); Eon aligner
  Arms: Clear aligner group
Device: Fixed pre-adjusted edgewise orthodontic appliance — Participants in this group will be treated with pre-adjusted fixed orthodontic appliances (Master Series®, American Orthodontics™, WI, USA). This system includes fixed brackets bonded on the labial surface of teeth and a sequence of progressively larger arch wires aimed at achieving alignment over time.
  Other Names: Fixed orthodontic appliance; Fixed labial braces; Conventional braces; Edgewise appliance; Fixed Appliance; Pre-adjusted Appliance; Straight-wire Appliance; Fixed Braces; Fixed Orthodontic Braces; Pre-adjusted Edgewise Bracket System; Straight-wire Bracket System; Fixed Multibracket Appliance; Fixed Straight-wire Technique
  Arms: Fixed labial braces group

SUMMARY:
The goal of this clinical trial is to compare between fixed labial braces and clear aligners for the straightening of moderately overlapped lower front teeth. The main questions it aims to answer are:

* Effect of treatment on gum health
* Which treatment achieves lower front teeth alignment faster in terms of alignment time and t number of visits required to the orthodontist
* How well it straightens teeth.

Participants will:

* Receive either labial braces or clear aligners as part of their orthodontic treatment.
* Come for regular follow-up visits every 4 to 6 weeks with the orthodontist till full straightening of the lower front teeth.
* Have a 3D scan of their teeth taken after their teeth are aligned along with a specialized x-ray of their head and jaw.

DETAILED DESCRIPTION:
The study is a randomized controlled trial aimed at comparing the efficiency, efficacy, periodontal and occlusal outcomes between two orthodontic treatment options: clear aligners and traditional fixed braces for patients with moderate crowding in the lower incisors.

Pre-treatment diagnostic records including clinical examination, intraoral scans, intraoral and extraoral photographs will be obtained for each participant.

To ensure that participants in both groups have similar levels of crowding severity and comparable dental health characteristics at the start of the study, randomization will be conducted in blocks. A total of forty participants (20 in each group) will be selected according to specific criteria designed to maintain this uniformity across both treatment groups.This study follows a parallel-group design and the participants will be randomly allocated into one of the two groups included in the study:

Intervention Groups:

* Group A - Fixed Labial Braces (Master Series®, American Orthodontics): In the traditional braces group, fixed metal brackets will be bonded to the lower teeth, and archwires will be used in a specific sequence designed to bring the teeth into alignment over time.
* Group B - Clear Aligners (EON Aligner): The clear aligner group will receive custom-fitted aligners created using a digital model of each participant's teeth. These aligners are removable, requiring patient adherence to wearing them for at least 22 hours daily.

Primary Outcomes:

1. Total alignment time
2. Clinical measures of periodontal status
3. Occlusal contact distribution
4. Efficacy of clear aligners Vs fixed appliances in alignment of lower anterior teeth

Secondary Outcomes:

1. Total number of scheduled routine appointments and additional emergency visits
2. Missed appointment rate
3. Number of refinements
4. Bracket/ attachment failure rate
5. Chair-side Time
6. Treatment Efficiency Index
7. BANA (Microbial-enzymatic N-benzoyl-DL-arginine-2-napthylamide) Score
8. Immunological Assay using ELISA
9. Patient's occlusal comfort level
10. Changes in mandibular incisor inclination
11. Changes in the mandibular arch form

Data will be analyzed using SPSS (Statistical Package for the Social Sciences) software, with statistical tests appropriate to the variable types (e.g., Mann-Whitney for group comparisons and Wilcoxon Signed-Rank test for time-related variables).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate lower crowding (Little's 4 to 6 mm), non-extraction treatment
* Age range: 13-45 years old
* Class I malocclusion
* Full permanent dentition
* No caries or periodontal disease

Exclusion Criteria:

* Extraction cases
* Patients with craniofacial syndromes, or cleft palate
* Patients with uncontrolled medical conditions or taking medication that can interfere with orthodontic tooth movement.
* Presence of extensive dental restorations in proximity to the gingival margin
* Presence of fixed bridges/crowns or partial dentures

Ages: 13 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Total alignment time | Through alignment, an average of 6 months
  The duration of treatment time (rounded to the nearest day) required to achieve full alignment of the mandibular incisors determined clinically as <1mm little's irregularity index, evaluated for both treatment groups. This information is to be extracted from participant notes into a data collection sheet designed specifically for this study.
Bleeding on probing | Baseline, after 3 months, and after 6 months
  Bleeding on probing as an indicator of tissue inflammatory response to bacterial pathogensis, using the Michigan Williams probe assigned a score of 0 - 3 for each site.
Occlusal contact surface area | Baseline, and after an average of 6 months, and after treatment an average of 1 year
  Occlusal contact surface area as measured by the T-scan device in terms of no. of pixels
Efficacy of clear aligners Vs fixed appliances in alignment of lower anterior teeth | Baseline, and after an average of 6 months
  Efficacy of clear aligners Vs fixed appliances in alignment of lower anterior teeth using Little's irregularity index
Symmetry of contact distribution | Baseline, and after an average of 6 months
  Symmetry of contact distribution as measured by the T-scan device.
Probing depth | Baseline, after 3 months, and after 6 months
  The distance measured from the base of the pocket to the most apical point on the gingival margin using the Michigan Williams probe.
Plaque index | Baseline, after 3 months, and after 6 months
  Plaque index to evaluate the level and rate of plaque formation on tooth surfaces
Gingival index | Baseline, after 3 months, and after 6 months
  Gingival index to determine the severity of gingival inflammation with a score from 0 - 3
Total treatment time | Through treatment, an average of 1 year
  The duration of treatment time (rounded to the nearest day) required to complete treatment, evaluated for both treatment groups. This information is to be extracted from participant notes into a data collection sheet designed specifically for this study.

SECONDARY OUTCOMES:
Total number of scheduled routine appointments and additional emergency visits | Through alignment, an average of 6 months
  The number of scheduled routine appointments required to achieve full mandibular incisor alignment and additional visits for emergencies as recorded in participants' notes and the data collection sheet.
Missed appointment rate | Through alignment, an average of 6 months
  The number of scheduled routine appointments that the patient failed to attend during the alignment phase of treatment as recorded in both participants' notes and the data collection sheet.
Number of refinements | Through alignment, an average of 6 months
  If any of the participants required a refinement scan prior to completion of leveling and alignment of the mandibular incisors, this would be recorded in both participants' notes and the data collection sheet
Bracket/ attachment failure rate | Through alignment, an average of 6 months
  Adverse events i.e., bracket failure rate in Group A and attachment failure rate in Group B were recorded in both participants' notes and the data collection sheet. The patient's provider noted in the clinical chart every bracket that had bond failure during the course of the study trial period. The brackets on the molar teeth were omitted. Brackets that debonded twice or more on the same tooth were counted only once. At the end of 180 days post-bonding, the percentage of broken brackets was calculated as: number of debonded brackets divided by the total number of teeth bonded (excluding molar teeth).
Chair side time | Through alignment, an average of 6 months
  The average time taken at the initial banding and bonding visit for the group A and the initial attachment bonding and aligner delivery visit for group B along with multiple routine mid-treatment appointments for both the groups during the alignment phase of treatment, as well as one emergency appointment for both measured using a digital stopwatch. The appointment times were rounded to the nearest minute with the total chair side time beginning when the patient sits on the chair and ending when they stood up to leave.
Treatment Efficiency Index | Through alignment, an average of 6 months
  The treatment efficiency index calculated by measuring the average Little's irregularity index before treatment and dividing it by the average treatment time in months/ days for alignment of the mandibular incisors.
BANA (Microbial-enzymatic N-benzoyl-DL-arginine-2-napthylamide) Score | Baseline, after 3 months, and after 6 months
  Microbiological index for the subgingival plaque
Immunological Assay using ELISA | Baseline, after 3 months, and after 6 months
  Immunological assay cytokine IL-1Beta in the gingival crevicular fluid
Patient's occlusal comfort level | Baseline, and after an average of 6 months, and after treatment an average of 1 year
  Patient's occlusal comfort level assessed by means of a Visual Analog Scale with a score from 0 - 10, 0 being least comfortable and 10 being most comfortable
Changes in mandibular incisor inclination | Baseline, and after an average of 6 months
  Changes in mandibular incisor inclination as measured on the lateral cephalogram
Changes in the mandibular arch form | Baseline, and after an average of 6 months
  Changes in the mandibular arch form as measured on the study model

CONTACTS AND LOCATIONS:
Overall Officials: Mais Medhat Sadek, BDS, MSc, PHD, Morth(RCSEd), Principal Investigator — University of Sharjah
Locations (1):
- University Dental Hospital Sharjah (UDHS_, Sharjah city, Emirate of Sharjah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available once the trial is finalized up to 3 years post recruitment
Access Criteria: Principle investigator and researchers will have access to all IPD collected throughout the trial once it has been depersonalized.

REFERENCES:
- [Background] Buschang PH, Shaw SG, Ross M, Crosby D, Campbell PM. Comparative time efficiency of aligner therapy and conventional edgewise braces. Angle Orthod. 2014 May;84(3):391-6. doi: 10.2319/062113-466. Epub 2013 Nov 18. PMID 24749702